CLINICAL TRIAL: NCT03791931
Title: Is Abnormal Cleavage Pattern of Embryos Associated With Different Oxidative Parameters Compared With That of Normally Cleaving Embryos? A Prospective Cohort Study
Brief Title: Cleavage Pattern of Embryos and Oxidative Parameters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Zofnat Wiener, Principal investigator, Carmel Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CMC 18-0087-CTIL
Record Dates: First submitted 2018-12-26; First posted 2019-01-03 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Other): Oxidative stress measurement in cleavage state embryos
  Interventions: Diagnostic Test: oxidative stress measurement

INTERVENTIONS:
Diagnostic Test: oxidative stress measurement — oxidative stress measurement

SUMMARY:
To investigate prospectively whether embryos with abnormal cleaving pattern have different oxidative parameters from normally cleaving embryos, and to analyze whether these parameters have an association with demographic, laboratory and clinical parameters including treatment outcome.

DETAILED DESCRIPTION:
To investigate prospectively whether embryos with abnormal cleaving pattern have different oxidative parameters from normally cleaving embryos, and to analyze whether these parameters have an association with demographic, laboratory and clinical parameters including treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing IVF for the treatment of infertility

Exclusion Criteria:

* Age <18 or >45 years old
* Patients with no embryos with direct cleavage

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-07-07 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
implantation rate | 1 year
  Implantation rate (positive BHCG)
clinical pregnancy rate | 1 year
  Clinical pregnancy as defined by appearance of gestational sac on ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Zofnat Wiener, MD, Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No